CLINICAL TRIAL: NCT07335315
Title: Evaluation of Intraoperative Contrast Enhanced Ultrasound for the Identification of Pituitary Adenoma in Cushing's Disease Compared to Other Pituitary Tumors
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: American Society of Head and Neck Radiology (Unknown); GE Healthcare (Industry); Lantheus Medical Imaging (Industry)
Responsible Party: Principal Investigator, Ian T. Mark, Principal Investigator, Mayo Clinic
Other Study IDs: 23-009009
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pituitary Adenoma; Cushing Disease
MeSH Terms: conditions — Pituitary Neoplasms; Pituitary ACTH Hypersecretion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Contrast: Patients who are scheduled for transsphenoidal surgical resection for Cushing disease or transsphenoidal resection for non-corticotroph adenomas.
  Interventions: Diagnostic Test: Contrast enhanced pituitary magnetic resonance imaging (MRI); Diagnostic Test: Contrast enhanced ultrasound
- Non-Contrast: Patients who are scheduled for a pituitary surgical procedure requiring an intra-operative ultrasound without contrast.
  Interventions: Diagnostic Test: Non-Contrast Ultrasound

INTERVENTIONS:
Diagnostic Test: Contrast enhanced pituitary magnetic resonance imaging (MRI) — Pre-operative contrast enhanced pituitary MRI and non-contrast intraoperative ultrasound.
  Groups: Contrast
Diagnostic Test: Contrast enhanced ultrasound — Contrast enhanced intraoperative ultrasound imaging with Definity microbubbles that will be activated per the manufacturer specification and administered as a bolus of 0.2 mL of perflutren lipid microsphere intravenously followed by a 10 mL flush of saline. The pituitary will be imaged in the transverse plane for 2 minutes following this bolus.
  A repeat injection of the same ultrasound contrast dose and saline flush will be performed, and the pituitary will be imaged in the sagittal plane for 2 minutes.
  Groups: Contrast
Diagnostic Test: Non-Contrast Ultrasound — Intra-operative ultrasound without contrast for pituitary adenomas and MRI
  Groups: Non-Contrast

SUMMARY:
This pilot and feasibility study aims to combine recent advances in ultrasound imaging, specifically an endonasal transducer array and contrast enhanced ultrasound, to offer an intraoperative image-guided solution for lesion-specific surgical resection to impact clinical outcome. Should this imaging approach help isolate specific lesions and prevent surgical resection of normal pituitary tissue in this first-in-humans study, then the results will provide clinical data for a much larger multi-center clinical trial.

ELIGIBILITY:
For Contrast Based Protocol:

Inclusion Criteria:

* Diagnosis of Cushing disease or required resection for non-corticotroph adenomas
* Agree to transsphenoidal resection.

Exclusion Criteria:

* Patients who are unable to consent (or if their legal guardian/representative decline to consent)
* Patients who have known or suspected hypersensitivity to microbubble contrast agents or its components such as polyethylene glycol (PEG).
* Women of child-bearing potential with a positive pregnancy test prior to procedure.
* Patients who have right to left, bi-directional, or transient right to left cardiac shunts.
* Patients who have hypersensitivity to perflutren.

For Non-Contrast Based Protocol:

Inclusion Criteria:

* Patients undergoing any pituitary surgery with the study designated neurosurgeons.
* Patients whose procedures require the use of an intra-operative BK ultrasound without contrast.

Exclusion Criteria:

• Patients who are unable to consent (or if their legal guardian/representative decline to consent)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a pituitary adenoma or lesion that will undergo transnasal surgery
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Scoring of non-contrast ultrasound images | Baseline
  Non-contrast ultrasound images will be evaluated by a board certified neuroradiologists with experience reviewing pituitary imaging. The ultrasound images will be scored on the identification, size, location, echogenicity, and enhancement of any potential pituitary lesions as well as a confidence level in identifying the adenoma (1-5 Likert scale) with 1 being non-diagnostic/poor and 5 being excellent/diagnostic quality.
Scoring of contrast-enhanced ultrasound images | Baseline
  Contrast-enhanced ultrasound images will be evaluated by a board certified neuroradiologists with experience reviewing pituitary imaging. The ultrasound images will be scored on the identification, size, location, echogenicity, and enhancement of any potential pituitary lesions as well as a confidence level in identifying the adenoma (1-5 Likert scale) with 1 being non-diagnostic/poor and 5 being excellent/diagnostic quality.
Scoring of pituitary MRI images | Baseline
  Preoperative Research Pituitary MRI images will be evaluated by a board certified neuroradiologists with experience reviewing pituitary imaging. The MRI images will be scored on the identification, size, location, echogenicity, and enhancement of any potential pituitary lesions as well as a confidence level in identifying the adenoma (1-5 Likert scale) with 1 being non-diagnostic/poor and 5 being excellent/diagnostic quality.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Mark, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No